CLINICAL TRIAL: NCT04701879
Title: Effect of Spinal Decompression Therapy With Core Stability Exercises in Radicular Chronic Low Back Pain
Brief Title: Spinal Decompression Therapy in Radicular Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aqua Medical Services (Pvt) Ltd (Industry)
Responsible Party: Principal Investigator, Mir Arif Hussain, Assistant professor, Aqua Medical Services (Pvt) Ltd
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/-00291 M.Umer
Record Dates: First submitted 2020-11-30; First posted 2021-01-08 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Radiculopathy Lumbar
Keywords: Physical therapy; Spinal decompression; Core stability exercises; Radiculopathy Lumbar
MeSH Terms: interventions — Laminectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spine decompression with core stability exercises (Active Comparator): Interventions in experimental group includes Hot pack, Spinal decompression therapy and core stability exercises
  Interventions: Other: Spine decompression with core stability exercises
- Spine decompression (Experimental): Intervention includesHot pack and spinal decompression therapy ..
  Interventions: Other: Spine decompression

INTERVENTIONS:
Other: Spine decompression with core stability exercises — * 50 minutes per session
  * Decompression with core stability on alternate days for 8 visits.
  Arms: Spine decompression with core stability exercises
Other: Spine decompression — 40 minutes per session
  -Decompression therapy on alternate days for 8 visits.
  Arms: Spine decompression

SUMMARY:
The study design was randomized control trial and sampling technique was lottery method. After inclusion and exclusion criteria, sample populations were divided into experimental (group A) and control group (group B). Spinal decompression therapy in combination with core stability exercises were given to experimental group as intervention while spinal decompression therapy given alone to the control group. Assessment was taken on after 1st session, 4th session and 8th session of physical therapy intervention. Data were entered and analyzed by SPSS version 21.

DETAILED DESCRIPTION:
Lower back pain is a common disorder that include any discomfort in the lumbar area below the origin of ribs and above the area of buttocks.Lower back pain with disability is 2nd most often reason for the wastage of time & money.Almost all people suffer from lower back pain at some age of their life .Both genders are effected equally by low back pain. The common problem of lower back pain are when you lift a heavy object prolonged unsupported sitting, accidents, sedentary life style. Sedentary life style could be the cause of low back pain usually when strenuous workout done on weekends as compared to minimal activities on week days. Lumbar area of the back hold and support the weight of the upper body and body do twisting and bending at this area. Specific or non-specific lower back pain is the classifications. Pain caused by any deformity, injury or any physical activity is called non-specific lower back pain.Non-specific lower back pain cannot be having any specific pathology, changes in behavior of movement pattern due to fear avoidance having bad postural control cause this non-specific pain.Lower back pain is one of the general health setbacks globally. It is the leading cause of people's absence from work and limits their activities.Prevalence and burden of low back pain increased with aging.Spinal decompression can create a opposite intradiscal pressure to promote led back of the herniated or bulging disc material and this oppsosity in the disc will cause influx of healing nutrients and other substances into the disc Core stability program improves functional status; reduce pain, increases quality of life and endurance of muscles in lumbar disk herniation patients.A strong core is important to the healthy spine. Abdominal muscle can help the back muscle supporting supine. If core muscle are weak, supine carry extra pressure on your back muscles. For this stabilizing and core exercises are important to strengthen back spine. By increasing endurance of these muscles core muscle should be strong. Core stability program improves functional status; reduce pain, increases quality of life and endurance of muscles in lumbar disk herniation patients.In 2008, a researcher found that stabilization exercises helpful in spinal rehabilitation to prevent from any sports injury. Another study by Hodges in 2003 stated that exercises for central muscle is an developing process; additional work necessary to purify and authenticate move forward, mainly with reference to understand the neurobiology of chronic pain.A study in 2011 on comparison between stabilization plan and Pilates technique for treating Low back pain. Their results showed that, Pereira technique is not is not helpful in get better back pain and function, in comparison with control and lumbar stabilization exercise groups.In exercise plan Mat and gym ball exercise for strength training and step box were used to develop an independent habit of exercise .these exercise plan intend to increase strength of muscle and decrease pain. As a main exercise walking is, safe, suitable and easy to decrease low back pain because it does not involve forceful and twisting forward flexion.

ELIGIBILITY:
Inclusion Criteria:

* Radicular low back pain with minimum 3 months of duration
* Both gender ( male and female)
* Age 20-60 years
* Limited Straight Leg Raise.

Exclusion Criteria:

* With marked bony and soft tissue disease.
* Less than 20 and more than 60 years of age.
* Patients who don't have MRI reports

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
The Oswestry Disability Index (ODI) | 0 Day
  The most reliable tool used by the clinicians to determine the functional disability of patients. Now days, the gold standard tool used for functional outcome of lower back is ODI.
The Oswestry Disability Index (ODI) | 4th Day
  The most reliable tool used by the clinicians to determine the functional disability of patients. Now days, the gold standard tool used for functional outcome of lower back is ODI.
The Oswestry Disability Index (ODI) | 8th Day
  The most reliable tool used by clinicians to determine the functional disability of patients. Nowadays, the gold standard tool used for the functional outcomes of the lower back is ODI.

OTHER OUTCOMES:
Numeric pain rating scale | 0 day, 4th day, 8th day
  The NPRS is used as an alternative tool of VAS in which the subject responds to the intensity of pain from 0 to 10. The total number of NPRS is 0 to 10 from which zero is considered as no pain, one to three is considered as mild pain, four to six considered as moderate pain and seven up to 10 considered as severe pain. the patient is guided to score the intensity of pain from zero to ten by own self.
Plank test | 0 day, 4th day, 8th day
  The test used to assess the strength of core muscles is known as plank test. It controls the endurance of the back/core stabilizing muscles. The starting position of the participants is to support the body by their elbows and forearm when off from the ground. The patient is guided to hold this position maximally. The test will be ended if the participants are unable to hold this position and time is noted by stopwatch. Total completed time will be the score to assess the core muscle strength.

CONTACTS AND LOCATIONS:
Overall Officials: Dr M.Umer Iqbal, MS, Principal Investigator — Shifa Tameer e milat University
Locations (1):
- Aqua research Center, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Borenstein DG. Chronic low back pain. Rheum Dis Clin North Am. 1996 Aug;22(3):439-56. doi: 10.1016/s0889-857x(05)70281-7. PMID 8844907
- [Background] Simpson AK, Cholewicki J, Grauer J. Chronic low back pain. Curr Pain Headache Rep. 2006 Dec;10(6):431-6. doi: 10.1007/s11916-006-0074-3. PMID 17087868
- [Background] Hoy D, Brooks P, Blyth F, Buchbinder R. The Epidemiology of low back pain. Best Pract Res Clin Rheumatol. 2010 Dec;24(6):769-81. doi: 10.1016/j.berh.2010.10.002. PMID 21665125
- [Background] McCaskey MA, Wirth B, Schuster-Amft C, de Bruin ED. Dynamic multi-segmental postural control in patients with chronic non-specific low back pain compared to pain-free controls: A cross-sectional study. PLoS One. 2018 Apr 10;13(4):e0194512. doi: 10.1371/journal.pone.0194512. eCollection 2018. PMID 29634749
- [Background] Hoy D, March L, Brooks P, Blyth F, Woolf A, Bain C, Williams G, Smith E, Vos T, Barendregt J, Murray C, Burstein R, Buchbinder R. The global burden of low back pain: estimates from the Global Burden of Disease 2010 study. Ann Rheum Dis. 2014 Jun;73(6):968-74. doi: 10.1136/annrheumdis-2013-204428. Epub 2014 Mar 24. PMID 24665116
- [Background] Murray CJ, Vos T, Lozano R, Naghavi M, Flaxman AD, Michaud C, Ezzati M, Shibuya K, Salomon JA, Abdalla S, Aboyans V, Abraham J, Ackerman I, Aggarwal R, Ahn SY, Ali MK, Alvarado M, Anderson HR, Anderson LM, Andrews KG, Atkinson C, Baddour LM, Bahalim AN, Barker-Collo S, Barrero LH, Bartels DH, Basanez MG, Baxter A, Bell ML, Benjamin EJ, Bennett D, Bernabe E, Bhalla K, Bhandari B, Bikbov B, Bin Abdulhak A, Birbeck G, Black JA, Blencowe H, Blore JD, Blyth F, Bolliger I, Bonaventure A, Boufous S, Bourne R, Boussinesq M, Braithwaite T, Brayne C, Bridgett L, Brooker S, Brooks P, Brugha TS, Bryan-Hancock C, Bucello C, Buchbinder R, Buckle G, Budke CM, Burch M, Burney P, Burstein R, Calabria B, Campbell B, Canter CE, Carabin H, Carapetis J, Carmona L, Cella C, Charlson F, Chen H, Cheng AT, Chou D, Chugh SS, Coffeng LE, Colan SD, Colquhoun S, Colson KE, Condon J, Connor MD, Cooper LT, Corriere M, Cortinovis M, de Vaccaro KC, Couser W, Cowie BC, Criqui MH, Cross M, Dabhadkar KC, Dahiya M, Dahodwala N, Damsere-Derry J, Danaei G, Davis A, De Leo D, Degenhardt L, Dellavalle R, Delossantos A, Denenberg J, Derrett S, Des Jarlais DC, Dharmaratne SD, Dherani M, Diaz-Torne C, Dolk H, Dorsey ER, Driscoll T, Duber H, Ebel B, Edmond K, Elbaz A, Ali SE, Erskine H, Erwin PJ, Espindola P, Ewoigbokhan SE, Farzadfar F, Feigin V, Felson DT, Ferrari A, Ferri CP, Fevre EM, Finucane MM, Flaxman S, Flood L, Foreman K, Forouzanfar MH, Fowkes FG, Fransen M, Freeman MK, Gabbe BJ, Gabriel SE, Gakidou E, Ganatra HA, Garcia B, Gaspari F, Gillum RF, Gmel G, Gonzalez-Medina D, Gosselin R, Grainger R, Grant B, Groeger J, Guillemin F, Gunnell D, Gupta R, Haagsma J, Hagan H, Halasa YA, Hall W, Haring D, Haro JM, Harrison JE, Havmoeller R, Hay RJ, Higashi H, Hill C, Hoen B, Hoffman H, Hotez PJ, Hoy D, Huang JJ, Ibeanusi SE, Jacobsen KH, James SL, Jarvis D, Jasrasaria R, Jayaraman S, Johns N, Jonas JB, Karthikeyan G, Kassebaum N, Kawakami N, Keren A, Khoo JP, King CH, Knowlton LM, Kobusingye O, Koranteng A, Krishnamurthi R, Laden F, Lalloo R, Laslett LL, Lathlean T, Leasher JL, Lee YY, Leigh J, Levinson D, Lim SS, Limb E, Lin JK, Lipnick M, Lipshultz SE, Liu W, Loane M, Ohno SL, Lyons R, Mabweijano J, MacIntyre MF, Malekzadeh R, Mallinger L, Manivannan S, Marcenes W, March L, Margolis DJ, Marks GB, Marks R, Matsumori A, Matzopoulos R, Mayosi BM, McAnulty JH, McDermott MM, McGill N, McGrath J, Medina-Mora ME, Meltzer M, Mensah GA, Merriman TR, Meyer AC, Miglioli V, Miller M, Miller TR, Mitchell PB, Mock C, Mocumbi AO, Moffitt TE, Mokdad AA, Monasta L, Montico M, Moradi-Lakeh M, Moran A, Morawska L, Mori R, Murdoch ME, Mwaniki MK, Naidoo K, Nair MN, Naldi L, Narayan KM, Nelson PK, Nelson RG, Nevitt MC, Newton CR, Nolte S, Norman P, Norman R, O'Donnell M, O'Hanlon S, Olives C, Omer SB, Ortblad K, Osborne R, Ozgediz D, Page A, Pahari B, Pandian JD, Rivero AP, Patten SB, Pearce N, Padilla RP, Perez-Ruiz F, Perico N, Pesudovs K, Phillips D, Phillips MR, Pierce K, Pion S, Polanczyk GV, Polinder S, Pope CA 3rd, Popova S, Porrini E, Pourmalek F, Prince M, Pullan RL, Ramaiah KD, Ranganathan D, Razavi H, Regan M, Rehm JT, Rein DB, Remuzzi G, Richardson K, Rivara FP, Roberts T, Robinson C, De Leon FR, Ronfani L, Room R, Rosenfeld LC, Rushton L, Sacco RL, Saha S, Sampson U, Sanchez-Riera L, Sanman E, Schwebel DC, Scott JG, Segui-Gomez M, Shahraz S, Shepard DS, Shin H, Shivakoti R, Singh D, Singh GM, Singh JA, Singleton J, Sleet DA, Sliwa K, Smith E, Smith JL, Stapelberg NJ, Steer A, Steiner T, Stolk WA, Stovner LJ, Sudfeld C, Syed S, Tamburlini G, Tavakkoli M, Taylor HR, Taylor JA, Taylor WJ, Thomas B, Thomson WM, Thurston GD, Tleyjeh IM, Tonelli M, Towbin JA, Truelsen T, Tsilimbaris MK, Ubeda C, Undurraga EA, van der Werf MJ, van Os J, Vavilala MS, Venketasubramanian N, Wang M, Wang W, Watt K, Weatherall DJ, Weinstock MA, Weintraub R, Weisskopf MG, Weissman MM, White RA, Whiteford H, Wiebe N, Wiersma ST, Wilkinson JD, Williams HC, Williams SR, Witt E, Wolfe F, Woolf AD, Wulf S, Yeh PH, Zaidi AK, Zheng ZJ, Zonies D, Lopez AD, AlMazroa MA, Memish ZA. Disability-adjusted life years (DALYs) for 291 diseases and injuries in 21 regions, 1990-2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2197-223. doi: 10.1016/S0140-6736(12)61689-4. PMID 23245608
- [Background] Apfel CC, Cakmakkaya OS, Martin W, Richmond C, Macario A, George E, Schaefer M, Pergolizzi JV. Restoration of disk height through non-surgical spinal decompression is associated with decreased discogenic low back pain: a retrospective cohort study. BMC Musculoskelet Disord. 2010 Jul 8;11:155. doi: 10.1186/1471-2474-11-155. PMID 20615252
- [Background] Choi J, Lee S, Hwangbo G. Influences of spinal decompression therapy and general traction therapy on the pain, disability, and straight leg raising of patients with intervertebral disc herniation. J Phys Ther Sci. 2015 Feb;27(2):481-3. doi: 10.1589/jpts.27.481. Epub 2015 Feb 17. PMID 25729196
- [Background] Akhtar MW, Karimi H, Gilani SA. Effectiveness of core stabilization exercises and routine exercise therapy in management of pain in chronic non-specific low back pain: A randomized controlled clinical trial. Pak J Med Sci. 2017 Jul-Aug;33(4):1002-1006. doi: 10.12669/pjms.334.12664. PMID 29067082
- [Background] Werners R, Pynsent PB, Bulstrode CJ. Randomized trial comparing interferential therapy with motorized lumbar traction and massage in the management of low back pain in a primary care setting. Spine (Phila Pa 1976). 1999 Aug 1;24(15):1579-84. doi: 10.1097/00007632-199908010-00012. PMID 10457578
- [Background] Macario A, Richmond C, Auster M, Pergolizzi JV. Treatment of 94 outpatients with chronic discogenic low back pain with the DRX9000: a retrospective chart review. Pain Pract. 2008 Jan-Feb;8(1):11-7. doi: 10.1111/j.1533-2500.2007.00167.x. PMID 18211590